CLINICAL TRIAL: NCT05019287
Title: Safety and Efficacy Study of Allogeneic Human Menstrual Blood Stem Cells Secretome to Treat Severe Covid-19 Patients, Clinical Trial Phase I&II
Brief Title: Menstrual Blood Stem Cells in Severe Covid-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avicenna Research Institute (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 990308-026; 99/3436 (Other Grant/Funding Number: Avicenna Research Institute)
Record Dates: First submitted 2021-07-03; First posted 2021-08-24 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Cytokine Storm
Keywords: mesenchymal stem cells; menstrual blood stem cell; secretome; covid-19
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: 1. Biological: allogeneic human menstrual blood stem cells secretome Intravenous injection of 5 ml menstrual blood stem cells secretome on day 1, day 2, day 3, day 4, and day 5, based on the routine treatment of COVID-19
  2. Other: Intravenous saline injection (Placebo) Intravenous injection of 5ml of 0.9% saline on day 1, day 2, day 3, day 4, and day 5, based on the routine treatment of COVID-19
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessments regarding clinical recovery will be conducted by the outcomes assessors blind to treatment allocation. Due to the nature of the intervention, staff cannot be blinded to allocation, but the participants are blind to the group to which they belong. An employee outside the research team will feed data into the computer in separate datasheets so that the outcomes assessors can analyses data without having access to information about the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menstrual blood stem cell secretome group (Experimental): Intravenous Allogeneic Menstrual Blood Stem Cells Secretome injection+Routine treatment
  Interventions: Biological: Allogeneic human menstrual blood stem cells secretome
- Control group (Placebo Comparator): Intravenous saline injection (Placebo)+Routine treatment
  Interventions: Other: Intravenous saline injection

INTERVENTIONS:
Biological: Allogeneic human menstrual blood stem cells secretome — This COVID-19 Study intervention consists of Intravenous Allogeneic human menstrual blood stem cell (MenSC) secretome injection in addition to standard care. The MenSC were characterized as CD90+, CD73+, CD105+, and CD45-based on multiparameter flow cytometry.
  Arms: Menstrual blood stem cell secretome group
Other: Intravenous saline injection — Intravenous saline injection in addition to standard care
  Arms: Control group

SUMMARY:
In this randomized controlled trial (RCT), severe cases of COVID-19 infection will be treated with secretome of menstrual blood stem cells. The improvement in the clinical, laboratory and radiological manifestations will be evaluated in treated patients compared with the control group.

DETAILED DESCRIPTION:
The devastating effect of severe acute respiratory syndrome coronavirus-2 (SARS COV-2) infection is caused by a robust cytokine storm that leads to lung tissue damage. Several studies have found that the severity of the disease is correlated with the release of excessive proinflammatory cytokines, such as IL-1, IL-6, IL-12, IFN-γ, and TNF-α, preferentially targeting lung tissue. This finding was confirmed by the high level of plasma cytokines found in the most severe COVID-19 patients associated with extensive lung damage. As a result, it is essential to find an effective treatment option to control the devastating cytokine storm of COVID-19 and regenerate the damaged lung. Although mesenchymal stem cells are a powerful tool for clinical applications, they have limits in terms of administration, safety, and variability of therapeutic response. It is interesting to note that the MSC secretome composed of cytokines, chemokines, growth factors, proteins, and extracellular vesicles could be a valid alternative to their use. It is not only easier to preserve, transfer and produce the secretome, but also safer to administer.

Previous studies reported that the hypoxic condition of MSCs could enhance the release of their active soluble molecules known as Secretome-MSCs (S-MSCs), such as IL-10 and TGF-β that useful in alleviating inflammation. Moreover, they could also increase the expression of growth factors such as VEGF and PDGF that accelerate lung injury improvement. These active molecules could potentially serve as a biological therapeutic agent for treating the severe SARS-CoV-2 infection. According to recent studies, we successfully isolated the S-MSCs from their culture medium using tangential flow filtration (TFF) strategy with several molecular weight cut-off category. This study investigated the clinical outcomes of severe COVID-19 patients with several comorbidities treated with S-MSCs in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose clinical and laboratory test results have a positive diagnosis of Covid-19.
* Patients who are willing to participate as subjects in the study by signing the informed content.
* Diagnosed with severe pneumonia of COVID: respiratory distress, RR >30 times/min; resting oxygen saturation of 90% or less; arterial partial pressure of oxygen / oxygen concentration ≤300mmHg; Pulmonary infiltration more than 50% in 24 to 48 hours
* SARS-CoV-2 nucleic acid test was positive.

Exclusion Criteria:

* History of drug reactions or allergies
* Pneumonia caused by bacteria, Mycoplasma, Chlamydia, Legionella, fungi, or other viruses
* Airway obstruction due to lung cancer or unknown factors
* Carcinoid syndrome
* History of epilepsy and long-term use of anticonvulsant drugs during the last 3 years
* History of long-term use of immunosuppressive drugs
* History of chronic respiratory illness that requires long-term oxygen therapy
* The patient is on blood or peritoneal dialysis
* Creatinine clearance <15 ml / min
* Moderate to severe liver disease (Child-Pugh score> 12)
* History of deep vein thrombosis (DVT) or pulmonary embolism over the past 3 years
* Being under ECMO or high-frequency oscillatory ventilation support
* Diagnostic of HIV, hepatitis B, and syphilis
* Pregnant or lactating women
* Lack of consciousness and inability to provide informed consent by the patient

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Adverse reactions incidence | Day 0 - 28
  The proportion of participants with treatment-related Adverse Event as assessed by CTCAE v5.0.
Time to clinical improvement | Day 0 - 28
  Days from administration of the Investigational Product for improvement

SECONDARY OUTCOMES:
Assessment of serum CRP (mg/L) levels | Days 0, 5, 10, 14, and 28
  To evaluate the anti-inflammatory effect of the proposed treatment an assessment of the inflammatory markers
Assessment of serum LDH (U/L) levels | Days 0, 5, 10, 14, and 28
  To evaluate the anti-inflammatory effect of the proposed treatment an assessment of the inflammatory markers
Assessment of serum Ferritin (ng/ml) levels | Days 0, 5, 10, 14, and 28
  To evaluate the anti-inflammatory effect of the proposed treatment an assessment of the inflammatory markers
Assessment of serum D-dimer (microgr/ml) levels | Days 0, 5, 10, 14, and 28
  To evaluate the anti-inflammatory effect of the proposed treatment an assessment of the inflammatory markers
Immunological changes on CD4+ T and CD8+ T | Days 0, 5, 10, 14, and 28
  Evaluate immune system improvement with flow cytometry to analyze patients' immune cells
Lung Involvement | Day 0 - 28
  Side effects measured by Chest Readiograph Side effects measured by Chest Readiograph
Changes in Inflammatory cytokine IL 6 | Days 0, 5, 10, 14, and 28
  To assess the anti-inflammatory effect of the proposed treatment an assessment of the levels of IL6 in plasma.
Changes in anti-Inflammatory cytokine IL10 | Days 0, 5, 10, 14, and 28
  To assess the anti-inflammatory effect of the proposed treatment an assessment of the levels of IL10 in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Mina Fathi Kazerooni, MD, PhD, Principal Investigator — Nanobiotechnology Research Center Avicenna Research Institute, ACECR, TEHRAN, IRAN; Ali Dehghan-Manshadi, MD, Study Chair — Department of Infectious Diseases and Tropical Medicine - Iranian Research Center for HIV/AIDS,TUMS; Samrand Fattah-Ghazi, MD, Study Director — Tehran University of Medical Science (TUMS); Somaieh Kazemnejad, PhD, Study Chair — Nanobiotechnology Research Center Avicenna Research Institute, ACECR, TEHRAN, IRAN
Locations (1):
- Avicenna Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fathi-Kazerooni M, Fattah-Ghazi S, Darzi M, Makarem J, Nasiri R, Salahshour F, Dehghan-Manshadi SA, Kazemnejad S. Safety and efficacy study of allogeneic human menstrual blood stromal cells secretome to treat severe COVID-19 patients: clinical trial phase I & II. Stem Cell Res Ther. 2022 Mar 7;13(1):96. doi: 10.1186/s13287-022-02771-w. PMID 35255966